CLINICAL TRIAL: NCT01686399
Title: A Sustainable Diet for Hadassah Employees
Brief Title: A Sustainable Diet for Hadassah Employees Workers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Ram Weiss, Associate Professor, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HMO 0645-11
Record Dates: First submitted 2012-09-09; First posted 2012-09-18 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Obesity; Physical Activity
Keywords: Sustainable diet; Health promotion; Obesity
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The study has a single arm (Experimental): The study has one arm The whole population of the campus will be exposed to the intervention. the effectiveness will be assessed using a random selection twice - before and after the intervention
  Interventions: Behavioral: Nutritional and Activity Promotion

INTERVENTIONS:
Behavioral: Nutritional and Activity Promotion — Multi disciplinary nutritional and behavioral messages to improve diet and activity levels

SUMMARY:
The aim of this protocol is to use a multidisciplinary approach to convey nutrition and activity messages to randomly selected Hadassah Medical Center employees. The intervention will be for one academic year and include frontal talks, email and internet focus group interactions, public demonstrations and a focused intervention within the hospital kitchen.

The outcomes are specific parameters of dietary modifications, degree of physical activity and health related perspectives. Outcomes will be recorded at baseline and by the end of the intervention ( one year).

DETAILED DESCRIPTION:
The participants will be selected randomly from the campus employees. They will be exposed to multiple levels of health promotion at the work place as well as via multiple media tools. Analysis will be performed at baseline by using multiple nutrition and health perception questionnaires. A second group from the employees will be selected for assessment of the same outcomes at the end of the year.

ELIGIBILITY:
Inclusion Criteria:

Hadassah medical center employees Age 21-67

-

Exclusion Criteria:

- Refusal to participate

Ages: 21 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Change in amount of fruit/vegetable consumption per day | one year
  Amount of fruit/vegetable consumption will be evaluated via questionnaires

SECONDARY OUTCOMES:
Amount of physical activity per week | one year
  Amount of physical activity will be assessed via questionnaires

OTHER OUTCOMES:
Amount of soft drinks consumed per day | one year
  The amount of soft drinks consumed per day will be assessed via questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Ram Weiss, MD PhD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem Region, Israel